CLINICAL TRIAL: NCT00489320
Title: An Observational Registry Using Drug Eluting Stents (DES) in Patients in a Real-World Setting (DEScover Registry).
Acronym: DESCOVER
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Other Study IDs: DESCOVER
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Diseases; Vascular Disease; Arterial Occlusive Disease; Arteriosclerosis; Atherosclerosis
Keywords: Coronary disease; Arteries; Atherosclerosis; Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Arterial Occlusive Diseases; Arteriosclerosis; Atherosclerosis; Coronary Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cypher Stent

SUMMARY:
The DEScover Registry is designed to observe the results of using Drug Eluting Stents (DES) in patients in a real-world setting. The stents being observed are not investigational, that is, they have been approved for use in the general population.

DETAILED DESCRIPTION:
The D.E.S.cover Registry is a prospective, multi-center, observational study. Consecutive patients undergoing PCI procedures will be asked to consent to participate in this study. For these patients, baseline, clinical and angiographic characteristics, as well as certain procedural and clinical events will be recorded using standardized case report forms. Outcomes will be assessed during hospitalization and at one, six and twelve months after discharge. Depending on results from the first year of follow-up, the study may be extended with an additional one or two years of follow-up.

The strategy for achieving the scientific objectives of the Registry is to document actual, real-world PCI practice and outcomes. Accordingly, the D.E.S.cover Registry does not specify treatment protocols, require any particular assignment of patients to treatment protocols, or in any other way require participating physicians to alter their practice patterns. Participating physicians are instructed to continue to treat all patients according to their own best clinical judgment, but to submit information on the parameters and outcomes of this treatment to the D.E.S.cover Registry database.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing percutaneous coronary intervention at an enrolling center by study investigators

Exclusion Criteria:

* Patient refusal or inability to provide written informed consent and/or HIPAA authorization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7759 (Actual)
Dates: Start 2004-12; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Williams, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Williams DO, Abbott JD, Kip KE; DEScover Investigators. Outcomes of 6906 patients undergoing percutaneous coronary intervention in the era of drug-eluting stents: report of the DEScover Registry. Circulation. 2006 Nov 14;114(20):2154-62. doi: 10.1161/CIRCULATIONAHA.106.667915. Epub 2006 Oct 23. PMID 17060386